CLINICAL TRIAL: NCT05486364
Title: A Study of Intermittent Photoplethysmography Based Rhythm Monitoring for Detection of Atrial Fibrillation Recurrence After Pulmonary Vein Isolation
Brief Title: DIGITal mOnitoring afTer Af abLation
Acronym: DIGITOTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Laurent Pison, Clinical professor, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Z-2021058
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Recurrent; PVI
Keywords: Atrial Fibrillation; PVI; Atrial ablation; pulmonary vein isolation; PPG; Photoplethysmography; Digital Health
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All subjects will receive both standard of care monitoring and digital rhythm monitoring using a PPG based smartphone application for AF recurrence after the PVI procedure.
  Interventions: Diagnostic Test: Digital Monitoring; Diagnostic Test: Standard of care

INTERVENTIONS:
Diagnostic Test: Digital Monitoring — Subjects will perform self-measurements with a PPG based smartphone application (FibriCheck™) to monitor for AF recurrence after the PVI procedure. One-minute measurements will be performed twice daily starting one month before the PVI procedure and continue up to 12 months after the procedure.
Diagnostic Test: Standard of care — Subjects will wear a 24-hour holter monitor at 3, 6 and 12 months after the PVI procedure. Additionally, outpatient cardiology clinic visits are organised at 6 weeks, 3 months and 12 months after the PVI procedure (including a 12-lead ECG and cardiologist consultation).

SUMMARY:
Recurrence of atrial fibrillation (AF) after a pulmonary vein isolation (PVI) procedure is frequent. Current follow up with Holter monitoring and electrocardiograms (ECG) during outpatient clinic consultations cover only short time stretches and require hospital visits. Mobile health solutions with rhythm monitoring using photoplethysmography (PPG) technology on a smartphone could extend rhythm monitoring time, while lowering hospital visits and cost. This study aims to compare the performance of a digital health solution using PPG technology on a smartphone versus the current standard of care to monitor for AF recurrence after a PVI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for an ablation procedure for AF, at least 4 weeks after the inclusion.
* Subject provides informed consent.
* Subject understands and agrees to comply with planned study procedures.
* Subject is able to perform measurements of the heart rhythm using the FibriCheck application at home.

Exclusion Criteria:

* Insufficient cognitive or comprehensive level of Dutch to participate to the trial.
* No access to a smartphone or unable to perform FibriCheck measurements at home.
* Pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
AF detection rate with PPG-monitoring vs standard of care monitoring after the blanking period in the first-year post AF ablation | 1 year

SECONDARY OUTCOMES:
Time to detection of AF after PVI (and after the blanking period) with PPG monitoring vs standard of care monitoring. | 1 year
The number and dispersion of PPG measurements needed to achieve similar sensitivity with intermittent one-minute PPG measurements compared to one 24h-Holter. | 1 year
Sensitivity, specificity and accuracy of PPG rhythm monitoring for AF detection during 24h-Holter monitoring on PPG measurement level. | 1 year
Proportion of confirmed symptom-rhythm correlations by PPG-monitoring vs standard care monitoring in patients who report symptoms on outpatient consultations. | 1 year
Predictive value of AF detection with PPG during blanking period for AF recurrence. | 1 year

OTHER OUTCOMES:
Patient compliance with PPG measurements | 1 year
Evaluation of AF-burden quantification by intermittent PPG measurements. | 1 year
Subanalysis of primary outcome 1 and secondary outcomes 1,2 and 3 | 1 year
  Excluding ECG measurements that were triggered by AF detection with PPG.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium